CLINICAL TRIAL: NCT02192853
Title: Plasma and Endothelial Activity of Dipeptidyl Peptidase 4 During Different Doses of Sitagliptin
Brief Title: Correlation Between Plasma- and Endothelial DPP-4 Activity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Emilie Skytte Andersen, Research student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-2-2012-149
Record Dates: First submitted 2014-01-04; First posted 2014-07-17 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus; Glucagon-like peptide 1; Dipeptidyl peptidase 4; Dipeptidyl peptidase 4 inhibitor; sitagliptin; Enzyme activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: intervention was blinded for the participant and the investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental): Patients with Type 2 Diabetes Mellitus and healthy control subjects are given tablets of sitagliptin in either a dosage of 25, 100 or 200 mg tablet in 3 different days.
  Interventions: Drug: sitagliptin
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sitagliptin — In randomized order:
  Day 1: tablet of 25 mg of sitagliptin + i.v. GLP-1 infusion Day 2: tablet of 100 mg of sitagliptin + i.v. GLP-1 infusion Day 3: tablet of 200 mg of sitagliptin + i.v. GLP-1 infusion
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — Day 4: placebo tablet
  Arms: placebo

SUMMARY:
The investigators want to estimate both the endothelial and the plasma activity of dipeptidyl peptidase 4 during different doses of sitagliptin in healthy subjects and patients with type 2 diabetes. Furthermore, the investigators want to investigate whether the current clinical dose of 100 mg of sitagliptin is sufficient to inhibit both the plasma and the endothelial activity of the enzyme dipeptidyl peptidase 4.

DETAILED DESCRIPTION:
The two incretin hormones glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP) are secreted from the intestinal L- and K- cells, respectively in response to ingestion of nutrients. The two hormones are able to lower blood glucose levels during high glucose levels - by the so called incretin effect. GIP and GLP-1 are both rapidly inactivated by the enzyme dipeptidyl peptidase 4 (DPP-4). The remaining metabolites are without insulinotropic effects. The effect of DPP-4 inhibitors used in treatment of type 2 diabetes relies on their impact on DPP-4 activity.

DPP-4 exists in a soluble form in plasma ad as a membrane-bound form in blood vessels and other tissues. The impact of DPP-4 inhibitors on DPP-4 activity has only been evaluated in plasma. We aim to investigate plasma and endothelial DPP-4 activity (i.e. whole-body DPP-4 activity) in patients with type 2 diabetes during different doses of the DPP-4 inhibitor sitagliptin.

Both healthy control subjects and patients with type 2 diabetes are subjected to 4 experimental days (in a randomized order) with continuous infusion of GLP-1 and pre-treatment with 25 mg sitagliptin, 100 mg sitagliptin, 200 mg sitagliptin and placebo, respectively. Afterwards, we are going to measure the whole-body DPP-4 activity by comparing plasma levels of active (intact) GLP-1 and total GLP-1, and relate to plasma DPP-4 activity.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians with diet and/or metformin treated patients with type 2 diabetes (diagnosed according to the criterias of the World Health Organization)
* Normal Hemoglobin
* Prior Informed Consent

Exclusion Criteria:

* Nephropathy
* Liver disease
* Inflammatory bowel disease
* Pregnancy

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Correlation between the total and intact GLP-1 hormone during different doses of sitagliptin measured as total area under the curve (tAUC) | GLP.1 total and GLP-1 intact will be calculated based on blood samples at time points: -40,-30,-20,-10,0,10,20,30,40,50,60,75,90,105,120,150,180,240,300,360 on all days

SECONDARY OUTCOMES:
Differences in serum-/plasma concentrations of GLP-1 measured as total Area under the curve (tAUC) | GLP-1 will be measured at time points(minutes): -40,-30,-20,-10,0,10,20,30,40,50,60,75,90,105,120,150,180,240,300,360 on all days
Differences in glucose measured as total Area under the curve (tAUC) | Glucose will be measured at time points(minutes): -40,-30,-20,-10,0,10,20,30,40,50,60,75,90,105,120,150,180,240,300,360 on all days
Differences in Insulin measured as total Area under the curve (tAUC) | Insulin will be measured at time points(minutes): -40,-30,-20,-10,0,10,20,30,40,50,60,75,90,105,120,150,180,240,300,360 on all days

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD PhD, Study Director — Gentofte Hospital; Tina Vilsbøll, MD DMSc, Study Chair — Gentofte Hospital; Asger Lund, MD, Study Chair — Gentofte Hospital; Camilla Andersen, Med.stud., Study Chair — Gentofte Hospital; Jens Juul Holst, MD DMSc, Study Chair — Institute of biomedical sciences, University of Copenhagen; Emilie Skytte Andersen, Med.stud., Principal Investigator — Gentofte Hospital
Locations (1):
- Diabetes Research Division, Department of Endocrinology, Gentofte Hospital, Hellerup, Denmark

REFERENCES:
- [Background] Deacon CF, Hughes TE, Holst JJ. Dipeptidyl peptidase IV inhibition potentiates the insulinotropic effect of glucagon-like peptide 1 in the anesthetized pig. Diabetes. 1998 May;47(5):764-9. doi: 10.2337/diabetes.47.5.764. PMID 9588448
- [Background] Holst JJ. The physiology of glucagon-like peptide 1. Physiol Rev. 2007 Oct;87(4):1409-39. doi: 10.1152/physrev.00034.2006. PMID 17928588
- [Background] Holst JJ, Vilsboll T, Deacon CF. The incretin system and its role in type 2 diabetes mellitus. Mol Cell Endocrinol. 2009 Jan 15;297(1-2):127-36. doi: 10.1016/j.mce.2008.08.012. Epub 2008 Aug 20. PMID 18786605
- [Background] Orskov C, Wettergren A, Holst JJ. Biological effects and metabolic rates of glucagonlike peptide-1 7-36 amide and glucagonlike peptide-1 7-37 in healthy subjects are indistinguishable. Diabetes. 1993 May;42(5):658-61. doi: 10.2337/diab.42.5.658. PMID 8482423
- [Background] Nauck MA, Heimesaat MM, Behle K, Holst JJ, Nauck MS, Ritzel R, Hufner M, Schmiegel WH. Effects of glucagon-like peptide 1 on counterregulatory hormone responses, cognitive functions, and insulin secretion during hyperinsulinemic, stepped hypoglycemic clamp experiments in healthy volunteers. J Clin Endocrinol Metab. 2002 Mar;87(3):1239-46. doi: 10.1210/jcem.87.3.8355. PMID 11889194
- [Background] Gutzwiller JP, Drewe J, Goke B, Schmidt H, Rohrer B, Lareida J, Beglinger C. Glucagon-like peptide-1 promotes satiety and reduces food intake in patients with diabetes mellitus type 2. Am J Physiol. 1999 May;276(5):R1541-4. doi: 10.1152/ajpregu.1999.276.5.R1541. PMID 10233049
- [Background] Vilsboll T, Krarup T, Madsbad S, Holst JJ. Both GLP-1 and GIP are insulinotropic at basal and postprandial glucose levels and contribute nearly equally to the incretin effect of a meal in healthy subjects. Regul Pept. 2003 Jul 15;114(2-3):115-21. doi: 10.1016/s0167-0115(03)00111-3. PMID 12832099
- [Background] Deacon CF. Circulation and degradation of GIP and GLP-1. Horm Metab Res. 2004 Nov-Dec;36(11-12):761-5. doi: 10.1055/s-2004-826160. PMID 15655705
- [Background] Herman GA, Stevens C, Van Dyck K, Bergman A, Yi B, De Smet M, Snyder K, Hilliard D, Tanen M, Tanaka W, Wang AQ, Zeng W, Musson D, Winchell G, Davies MJ, Ramael S, Gottesdiener KM, Wagner JA. Pharmacokinetics and pharmacodynamics of sitagliptin, an inhibitor of dipeptidyl peptidase IV, in healthy subjects: results from two randomized, double-blind, placebo-controlled studies with single oral doses. Clin Pharmacol Ther. 2005 Dec;78(6):675-88. doi: 10.1016/j.clpt.2005.09.002. PMID 16338283